CLINICAL TRIAL: NCT00407901
Title: Functional Assessment Questionnaire for the Visually Challenged: Proposed Model to Quantitatively Measure the Functional Level of Individuals Who Are Legally Blind
Brief Title: Functional Assessment Questionnaire for the Visually Challenged
Status: Completed | Type: Observational
Sponsor: George Washington University (Other)
Responsible Party: Dr. Craig Geist, M.D., M.S., The George Washington University University Medical Faculty Associates
Other Study IDs: GWUIRB#120526
Record Dates: First submitted 2006-12-01; First posted 2006-12-05 (Estimated); Last update posted 2008-01-18 (Estimated); Status verified 2008-01

CONDITIONS: Blindness, Legal
Keywords: Visually Challenged; Legally Blind; Functional Assessment Questionnaire; Low Functioning; High Functioning
MeSH Terms: conditions — Blindness

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A, B: A: High functioning visually challenged (legally blind) B: Low-functioning visually challenged (legally blind)

SUMMARY:
The purpose of this research is to evaluate how accurately a proposed "Functionality Assessment Questionnaire" measures the differences between low-functioning and high-functioning visually challenged individuals who are legally blind.

DETAILED DESCRIPTION:
The specific aim of this research is to establish the scientific validity of an evaluation assessment tool that will measure the functional level of the visually challenged population. For this study a quantitative, self-evaluation tool has been designed to assess the functional skills at performing a variety of activities. It is called the Functional Assessment Questionnaire. The questionnaire is an innovative approach to measuring the level of these functional skills. It also includes critical benchmarks of real-world success that are not considered in assessing functional levels of the visually challenged, but are measures of evidence-based outcomes. It is a comprehensive measurement tool covering many areas of daily living, including:

1. Education Level
2. Employment Level
3. Income Level
4. Personal Living Skills
5. Kitchen Skills
6. Mobility Level
7. Reading/Writing Skills
8. Oral Communication Skills
9. Social Skills
10. Technology Level
11. Financial Management Skills
12. Recreation Skills
13. Organizational Skills
14. Independence Level

Each of these categories include a progressive scale of 10 activities, 1 being the lowest level of functionality and 10 being the highest level of functionality. Most of the categories are easily self-evaluated, though some will require one-on-one discussion with the test administrator. At the completion of the Functional Assessment Questionnaire, a functionality score, ranging between 14 and 140 is tabulated for each individual.

In order to maintain scientific integrity of the Functional Assessment Questionnaire, certain non-identifiable information will be collected on each human subject. This information includes:

1. Age
2. Sex
3. Visual Acuity (BCVA)
4. Peripheral Field
5. Diagnosed Eye Condition

Comparative statistical analysis will be performed with the Functional Assessment Questionnaire results and the widely used SF-36 (36-Item Short Form Health Survey Instrument) and NEI-VFQ-25 with Appendix (National Eye Institute/Visual Function Questionnaire-25) questionnaires. The goal will be to check which questionnaire is more sensitive and accurate in measuring functional level outcomes both prior to (low-functioning individuals) and after (high functioning individuals) vision rehabilitation program participation.

ELIGIBILITY:
Inclusion Criteria:

* Between ages of 18 and 80.
* Capacity to complete the informed consent process
* Legally blind (best corrected visual acuity of 20/200 or greater, and/or vision field of 20 degrees or less).
* Long-term or short-term blindness with no or minimal vision rehabilitation. (These will be considered low-functioning subjects). or
* Legally blind with extensive vision rehabilitation, independent and self-sufficient. (These will be considered high-functioning subjects).

Exclusion Criteria:

* Patients who have incapacitating physical and mental challenges other than vision loss.
* Patients who are not legally blind.
* Patients who have had some vision rehabilitation, thus falling in between a high-functioning and low-functioning category.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 30 legally blind individuals. Between 12-15 individuals will be categorized as poor or low-functioning, and the same number of subjects that are categorized as high-functioning.
  The factors that will establish high-functioning abilities will be outward skills in adapting to vision loss, such as:
  1. Employment in mainstream job market
  2. Extensive vision rehabilitation
  3. Inclusion into mainstream society
  4. Success in real world
  5. Demonstrated ability to live independently, shop, cook, clean, pay bills, and move around safely without assistance.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2006-04; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Geist, M.D., M.S., Principal Investigator — George Washington University

REFERENCES:
- [Result] Lingebach D, Olszowy R, Zollman R and Geist CE. Functional Assessment Questionaire for Low Vision. Abstract. Envision Conference, Kansas City, September 22-23, 2006 Poster Session.